CLINICAL TRIAL: NCT06583746
Title: Lower Extremity Evaluation in Children With Diparetic Cerebral Palsy According to ICF Perspective
Status: Completed | Type: Observational
Sponsor: Acıbadem Atunizade Hospital (Other)
Responsible Party: Principal Investigator, Ilayda Sozeri, Pediatric Physiotherapist, Acıbadem Atunizade Hospital
Other Study IDs: IlaydaS
Record Dates: First submitted 2024-09-02; First posted 2024-09-04 (Actual); Last update posted 2024-09-04 (Actual); Status verified 2024-09

CONDITIONS: Diparesis; Cerebral Palsy; Diplegic Cerebral Palsy; Lower Extremity Paresis
Keywords: Diparetic Cerebral Palsy; Lower extremity; International Classification of Function; Body structure and function; Activity; Participation
MeSH Terms: conditions — Cerebral Palsy; Paresis; Motor Activity

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Lower extremity evaluation of children with DCP within the framework of ICF: 30 children with DCP were included. The lower extremity evaluations of these cases were made according to ICF. Modified Ashworth Scale (MAS) was used for body structure and functions, Gillette Functional Assessment Questionnaire (FAQ) was used for activity and Pediatric Functional Independence Measure (WeeFIM) was used for participation.
  Interventions: Other: Group1

INTERVENTIONS:
Other: Group1 — 30 children with DCP were included. The lower extremity evaluations of these cases were made according to ICF. Modified Ashworth Scale (MAS) was used for body structure and functions, Gillette Functional Assessment Questionnaire (FAQ) was used for activity and Pediatric Functional Independence Measure (WeeFIM) was used for participation.

SUMMARY:
Cerebral palsy (CP); is the most common neurodevelopmental disorder seen in childhood, characterized by permanent motor dysfunctions that develop due to brain damage occurring before birth, during birth, or in early childhood.

The most common type is spastic type CP with a prevalence rate of 70-80%. Spastic type CP is divided into three groups as diparetic (38%), hemiparetic (39%) and quadriparetic (23%). In diparetic cerebral palsy (DCP); lower extremity involvement is more pronounced than upper extremity involvement. Typically; weakness in the trunk, postural and antigravity muscles, functional and/or structural asymmetry between both lower extremities are seen and this condition is closely related to impaired static and/or dynamic balance, decreased postural control, decreased functional performance, and low participation rate in activities.

The ICF (International Classification of Functioning, Disability, and Health) was developed by the World Health Organization in 2001 and is a comprehensive model that evaluates health status not only through the presence of diseases and disorders but also through various dimensions such as functionality, environmental, and personal factors. The ICF model includes five main components to evaluate an individual's functionality and disability: body structure and functions, activity, participation, environmental and personal factors. In recent years, functional abilities, including social participation, have increasingly become the focus of research in children with CP.

DETAILED DESCRIPTION:
It's an observational study.

Purpose of the study: The increase in tone seen in the lower extremities in children with diparetic cerebral palsy (DCP) may adversely affect the activity and participation of children. Our study aim is to evaluate lower extremities in children with DCP according to ICF perspective.

A total of 30 cases, 15 females (50%) and 15 males (50%), aged between 3 and 13 years (mean: 5.8), who were admitted to the Pediatric Rehabilitation Department of Acıbadem Altunizade Hospital with the diagnosis of DCP between 2019 and 2022, were included in this cross-sectional study.

* What should the rehabilitation program for children with DCP include?
* What should we consider when evaluating children with DCP?

The lower extremity evaluations of these cases were made according to ICF. Modified Ashworth Scale (MAS) was used for body structure and functions, Gillette Functional Assessment Questionnaire (FAQ) was used for activity, and Pediatric Functional Independence Measure (WeeFIM) was used for participation

ELIGIBILITY:
Inclusion Criteria:

* Between 3-13 years old,
* Diagnosis of diparetic cerebral palsy,
* Participants and/or parents willing to participate in the study voluntarily.

Exclusion Criteria:

* Having different types of CP such as dyskinetic, mixed, ataxic types other than spastic type,
* Having spastic quadriparetic or hemiparetic type CP,
* Having received Botulinum Toxin injections to the lower extremities within the last 6 months.

Ages: 3 Years to 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children diagnosed with diparetic cerebral palsy between the ages of 3 and 13 were included.
Sampling Method: Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2002-01-01 (Actual); Primary Completion 2022-01-31 (Actual); Study Completion 2022-01-31 (Actual)

PRIMARY OUTCOMES:
Modified Ashworth Scale (MAS) | baseline
  It is a 6-point scale used to describe the resistance of the muscle to passive movement and the ease with which the joint can be moved within the available range. It is frequently used in clinical settings. It is quite practical to evaluate and interpret.
Gillette Functional Walking Assessment Questionnaire (FAQ) | baseline
  It is a measurement tool used to evaluate walking ability and functional mobility in children. This questionnaire was developed specifically to evaluate the walking functions of children with cerebral palsy and other neuromuscular disorders. Developed at Gillette Children's Hospital, this questionnaire aims to rate children's walking abilities in different environments. It scores children's walking skills on a scale of 1-10.
Pediatric Functional Independence Scale (WeeFIM) | baseline
  The WeeFIM scale is a tool used to assess children's independence levels and functional abilities. It was developed to objectively assess children's independence levels and whether they need assistance with daily living activities. The scale consists of 6 main headings and 18 subheadings. These subheadings evaluate areas such as self-care (feeding, dressing, toilet use), sphincter control, transfers (e.g. bed, chair), movement (walking, wheelchair use), communication and social cognition (problem solving, memory). Scoring ranges from 1 to 7, with the highest score being 126. As the score increases, assistance decreases and independence increases.

CONTACTS AND LOCATIONS:
Locations (1):
- Acıbadem Altunizade Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be made available to other researchers.